CLINICAL TRIAL: NCT00285961
Title: Evaluation of Cork Splint Materials Instead of Plaster Splint for Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: René Verdonk, University Ghent
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003/364
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-02

CONDITIONS: Wrist Fractures; Forearm Fractures; Elbow Fractures; Ankle Fractures; Foot Fractures; Wounds and Injuries
Keywords: Fractures of the wrist, forearm, elbow, ankle, foot; Distortions of the wrist, elbow, ankle; Wounds without tendon injuries
MeSH Terms: conditions — Wrist Fractures; Elbow Fractures; Ankle Fractures; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Cork splint materials (instead of plaster splint)

SUMMARY:
This is an evaluation of the functionality and added value of cork splint materials instead of a plaster splint for children (3-11 years old).

ELIGIBILITY:
Inclusion Criteria:

* Fractures of the wrist, forearm, elbow, ankle, foot
* Distortions of the wrist, elbow, ankle
* Wounds without tendon injuries

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Functionality
Added value

CONTACTS AND LOCATIONS:
Overall Officials: Rene Verdonk, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be